CLINICAL TRIAL: NCT03782441
Title: A Pilot Study of a Novel Non-invasive Glucose Monitoring Device
Brief Title: Study of a Novel Non-invasive Glucose Monitoring Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RSP Systems A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: RSP-19
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2019-12

CONDITIONS: Diabetes Mellitus
Keywords: Non-invasive glucose monitoring; Raman spectroscopy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RSP-19 (Experimental): Subjects will perform daily measurements on the IMD (Prototype 0.5) for 42 days.
  Interventions: Device: Prototype 0.5

INTERVENTIONS:
Device: Prototype 0.5 — Investigational Medical Device collecting spectral Raman data from tissue

SUMMARY:
This explorative clinical study has been launched to collect spectral Raman data paired with validated glucose reference values in diabetic patients.

DETAILED DESCRIPTION:
The Investigational Medical Device (IMD) for this investigation is the Prototype 0.5 (P0.5) developed and manufactured by RSP Systems (RSP). The device is intended for non-invasive interstitial intermittent glucose monitoring in persons (age 18 and older) with diabetes. The technology relies on the well-established capacities of Raman spectroscopy for directly detecting glucose subcutaneously. The Raman spectroscopy physical principle relies on the fact that when laser light of a given wavelength interferes with a molecule, a small fraction of the incident light will interact with the vibrational states of the molecule, causing the photons to lose a portion of their energy which will change the wavelength of the light. The scattered light will be collected by the optical probe head and analyzed with advanced algorithms to correlate the signal to glucose concentrations. Data collected from the IMD will be paired with validated glucose reference values collected by the finger sticking method.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥18 years of age
* Diagnosed with diabetes, all types except gestational diabetes
* HbA1c distribution > 60 mmol/mol at baseline visit
* Skin phototype 1-4
* Willing to perform a minimum of 8 finger sticks during each day of home-based measurements and 30 finger sticks at the two in-clinic study days
* Subject has a wireless internet connection at home to be used in the study

Exclusion Criteria:

* For female subjects: Pregnancy or subject is attempting to conceive or not willing and able to practice birth control during the study duration
* For female subjects: Breastfeeding
* Subject currently participating in another study
* Subject not able to understand and read Danish
* In investigator's opinion, subject is not able to follow instructions provided and as specified in the protocol
* Subject not able to hold hand/arm steady (including tremors and Parkinson's Disease)
* Reduced circulation in right hand evaluated by Allen's test
* Extensive skin changes, tattoos or diseases on right hand thenar (probe application site)
* Known allergy to medical grade alcohol used to clean the skin
* Medical history or any condition that may, in the opinion of the investigator compromise the subject's ability to participate
* Comorbidity or concomitant medical condition which, in the opinion of the Investigator, could interfere with the study or present a risk to the safety or welfare of the subject or study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Measurement accuracy of IMD | 4 months
  Accuracy of measurements performed on the IMD will be evaluated by data from subjects. Data will be analyzed by Mean Absolute Relative Difference (MARD) and Inter Subject Unified Performance (ISUP)
Safety evaluation: paucity of adverse events | 4 months
  Safety of the IMD will be evaluated in a descriptive manner by the paucity of adverse events reported during the clinical study

SECONDARY OUTCOMES:
Device deficiency | 4 months
  Description of device deficiencies will be listed. Deficiencies will be reported during the clinical study.
Device usability | 4 months
  The use of the device by the subjects will be evaluated by means of questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Sanne Fisker, Principal Investigator — Steno Diabetes Center, Aarhus University Hospital
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No